CLINICAL TRIAL: NCT00790725
Title: Proportional Assist Ventilation vs. Pressure Support Ventilation in the Management of Patients Referred to a Respiratory Acute Care Unit
Brief Title: Proportional Assist Ventilation vs Pressure Support Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient population in RACU has changed significantly, we can not find potential subjects to recruit. The enrollment rate has reached zero.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Professor of Anesthesia, Director of Respiratory Care Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001377
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAV (Other): Proportional Assist Ventilation will be used as a mechanical ventilation method for randomized patients in RACU
  Interventions: Other: Proportional Assist Ventilation
- PS (Other): Pressure Support Ventilation will be used as a mechanical ventilation method for randomized patients in RACU
  Interventions: Other: Pressure Support Ventilation

INTERVENTIONS:
Other: Proportional Assist Ventilation — Proportional Assist Ventilation will be used to ventilate the patients.
  Arms: PAV
Other: Pressure Support Ventilation — Pressure Support ventilation will be used to ventilate the patients.
  Arms: PS

SUMMARY:
In this study, we want to compare two different kinds of artificial ventilation to see if one encourages faster weaning from breathing support and if one provides better sleep quality. These artificial ventilation types are:

1. Pressure support ventilation; the standard ventilation that we use for the patients in the Respiratory Acute Care Unit. Pressure support ventilation ventilators use constant air pressure to assist patients with their breathing.
2. Proportional assist ventilation; a newer way of helping people with their breathing. The air pressure provided by proportional assist ventilation ventilators varies with the size of the breath that a person takes.

ELIGIBILITY:
Inclusion Criteria:

* Tracheotomized or endotracheally intubated and mechanically ventilated patients transferred or scheduled to be transferred to the RACU.
* Age 18 years or older.

Exclusion Criteria:

* Patients who are weaned from ventilatory support within the first 72 hours of transfer to the RACU. Even though these patients had been randomized, they will be excluded. They will be considered in the intention to treat analysis but the final outcome analysis will be performed after their exclusion.
* High spinal cord injury
* Immunosuppressed patients receiving chemotherapy or radiation therapy (< 2 months after chemotherapy or radiation therapy).
* Neuromuscular/ neurological disease of a progressive nature resulting in chronic ventilator dependence.
* High risk of mortality within 3 months (severe neurological damage and cancer patients in terminal stages of the disease).
* Patients unable to trigger the ventilator for any reason.
* Any patient who is not considered a candidate for weaning from ventilatory support
* Patients consented for another interventional study.
* Patients requiring more than 30 days to wean once randomized will be excluded. They will be considered in the intention to treat analysis but the final outcome analysis will be performed after their exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Length of time mechanically ventilated in the RACU | 30 days

SECONDARY OUTCOMES:
Sleep quality | 48 hours
Inflammatory mediator levels | 30 days
Hospital mortality | 30 days
60 day mortality | 60 days
180 day mortality | 180 days
365 day mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States